CLINICAL TRIAL: NCT00955162
Title: A Multicentre, Randomised, Open-label, Active-controlled Trial of the Effectiveness of Buprenorphine/Naloxone in Reducing Intravenous Buprenorphine Misuse in France
Brief Title: Effectiveness of Buprenorphine/Naloxone in Reducing Intravenous Buprenorphine Misuse in France ("RIME")
Acronym: RIME
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BU0902
Record Dates: First submitted 2009-08-05; First posted 2009-08-07 (Estimated); Last update posted 2012-11-30 (Estimated); Status verified 2010-01

CONDITIONS: Opioid Dependency
Keywords: Substance Abuse, Intravenous; Buprenorphine
MeSH Terms: conditions — Substance Abuse, Intravenous | interventions — Buprenorphine; Naloxone; Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subutex (Active Comparator)
  Interventions: Drug: Buprenorphine (Subutex)
- Suboxone (Experimental)
  Interventions: Drug: Buprenorphine/naloxone (Suboxone)

INTERVENTIONS:
Drug: Buprenorphine (Subutex) — Sublingual tablet
  Other Names: Subutex
  Arms: Subutex
Drug: Buprenorphine/naloxone (Suboxone) — Sublingual tablet
  Other Names: Suboxone
  Arms: Suboxone

SUMMARY:
Patients who admit to using buprenorphine by the intravenous route will be randomized to either Subutex or Suboxone and be followed up for 3 months to determine if there is less injection with Suboxone than with Subutex based primarily on patient diaries.

Patients randomized to Suboxone may continue to receive the product for a further 9 months at their request and will be monitored at 3 month intervals.

Patients will receive a payment for the inconvenience of keeping a daily diary and to cover their travel expenses.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female opioid-dependent outpatient aged 18 years or older,
2. Women of childbearing potential must have a negative urine pregnancy test result at the Inclusion Visit (test under supervision of the investigator or designee),
3. Women of childbearing potential must use an effective birth control method. Women of non-childbearing potential must be postmenopausal or must be surgically sterile (hysterectomy and/or bilateral oophorectomy),
4. On buprenorphine (Subutex® or generic buprenorphine) maintenance therapy at a minimum daily dose of 2 mg for at least 3 months prior to inclusion,
5. Declaring buprenorphine intravenous misuse at least four times/week and showing needle marks,
6. Willing to stop or reduce buprenorphine intravenous misuse,
7. Having received oral and written information about the trial, and provided written informed consent prior to admission to this trial.

Exclusion Criteria:

1. Pregnancy or breast-feeding,
2. Contraindication or history of hypersensitivity to buprenorphine, naloxone or to any excipient of Suboxone® or Subutex®,
3. Any medical or psychiatric condition which in the opinion of the investigator would make participation difficult or unsafe,
4. Participating in another trial,
5. Patients in the exclusion period of the "Fichier National des personnes qui se prêtent à des recherches biomédicales" (National Index of persons participating in biomedical researches, or National Index of volunteers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
number of study drug injections per week | 1 week

SECONDARY OUTCOMES:
Addiction severity | 3 months
Withdrawal severity | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Didier TOUZEAU, MD, Principal Investigator — Hôpital Paul Guiraud, Bagneux
Locations (20):
- France (20):
  - Csst Antibes, Antibes
  - Hopital Paul Guiraud, Bagneux
  - Cssa Bizia, Bayonne
  - Centre Carreire , CH Charles Perrens, Bordeaux
  - CHU de Clermont-Ferrand, Centre Méthadone, Clermont-Ferrand
  - Service d'addictologie, Hopital de Dole, Dole
  - CSST NAUTILIA (Ex Alinea), Le Havre
  - CSST Le Cèdre Bleu, Lille
  - Centre Hospitalier Esquirol - Intersecteur, Regional Soins en Addictologie, Limoges
  - Centre Baudelaire, Metz
  - Csst de Montauban, Montauban
  - CSST Centre Hospitalier, Nice
  - CSST Logos, Nîmes
  - Hôpital Caremeau, Nîmes
  - Csst Espace Murger, Paris
  - Hôpital Saint Anne, Paris
  - Centre L'Envol (Csst), Rennes
  - Centre Baudelaire, Thionville
  - Hopital Joseph Ducuing, Toulouse
  - CSST Centre Port Bretagne CH Charles Perrens, Tours